CLINICAL TRIAL: NCT06478030
Title: Combined Screening for Gastrointestinal Tumors
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Fenghua District People's Hospital, Ningbo City (Unknown); Fenghua District Traditional Chinese Medicine Hospital, Ningbo City (Unknown); Xikou Hospital in Fenghua District, Ningbo City (Unknown); Yongkang Traditional Chinese Medicine Hospital (Unknown); Hangzhou Medical College (Other)
Responsible Party: Principal Investigator, Xiangdong Cheng, Chief physician, Zhejiang Cancer Hospital
Other Study IDs: IRB-2023-890
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Gastrointestinal Tumors
MeSH Terms: conditions — Digestive System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — stool, urine, blood, tongue coating, saliva, gastric juice, and fresh tissue (gastric mucosa tissue and/or intestinal polyp tissue).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Screening cohort: Healthy participants aged 40-74 years from designated communities.
  Interventions: Diagnostic Test: questionnaire, Helicobacter pylori (H. pylori) test, fecal immunochemical test (FIT)

INTERVENTIONS:
Diagnostic Test: questionnaire, Helicobacter pylori (H. pylori) test, fecal immunochemical test (FIT) — The questionnaire covers nine aspects: basic information of the participants, symptoms and previous examinations, medical history and surgical history, medication history, smoking history, alcohol consumption history, dietary habits, physical exercise, and family history.

SUMMARY:
All participants are required to complete a questionnaire, a Helicobacter pylori (H. pylori) test, and a fecal immunochemical test (FIT). The questionnaire covers nine aspects: basic information of the participants, symptoms and previous examinations, medical history and surgical history, medication history, smoking history, alcohol consumption history, dietary habits, physical exercise, and family history. After quality control, the data is entered by staff into the Zhejiang Province Cancer Screening Information Platform. Risk assessments are performed based on the data collected and high-risk individuals are recommended for clinical screening. Additionally, tongue image, stool, urine, blood, tongue coating, saliva, gastric juice, and fresh tissue (gastric mucosa tissue and/or intestinal polyp tissue) samples are collected from all participants undergoing clinical screening.

Participants are required to complete at least one passive follow-up annually. Active follow-ups are conducted for those with positive screening results to ensure timely completion of endoscopic examinations. For those who have not undergone endoscopic examinations despite positive screening results, health education is provided, and they are mobilized at least four times within one month to complete endoscopic examinations. For participants diagnosed and treated for precancerous lesions and tumors, diagnostic and treatment data must be collected, and they are encouraged to follow up as per medical advice. Both active and passive follow-up results must be recorded in the screening follow-up information record form and reported to the Zhejiang Province Cancer Screening Information Platform.

This is a government collaboration project. All subjects will also be followed by record linkage to Cancer Register and Population Register.

ELIGIBILITY:
Inclusion Criteria:

* Subject residents from Zhejiang Province.
* Subject is able to comprehend, sign, and date the written informed consent document to participate in the study.
* Subject has psychical condition and well consciousness, and also accept and cooperate with the follow-up of this study.

Exclusion Criteria:

* Subject has heavy cardiovascular, liver or kidney disease.
* Subject is already suffering from malignant tumors of the digestive tract.
* Subject has severe intellectual disabilities or language communication barriers.
* Subject has had gastrointestinal endoscopy in the past year.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population data obtained from local government departments is used to identify eligible participants. From this pool, individuals who meet the criteria are selected, and their names along with basic information are recorded.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal cancers detection, incidence and mortality | 5 years
  Gastrointestinal cancers detection through endoscopies, and gastrointestinal cancers incidence and mortality with long-term follow-up.

SECONDARY OUTCOMES:
Early diagnosis of gastrointestinal cancers | 5 years
  Early diagnosis of gastrointestinal cancers using different strategies.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Yongkang City, Jinhua, Zhejiang
  - Fenghua District, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No
Not provided